CLINICAL TRIAL: NCT04961216
Title: Effectiveness of an Online Programme to Tackle Individual's Meat Intake Through SElf-regulation (OPTIMISE): A Randomised Controlled Trial
Brief Title: The OPTIMISE Intervention for Reducing Meat Consumption in UK Adult Meat-eaters
Acronym: OPTIMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, ProfessorSusanJebb, Professor of Diet and Population Health, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R71398/RE002
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Diet Habit
Keywords: self-regulation; self-monitoring; goal-setting; meat reduction; multi-component intervention
MeSH Terms: conditions — Feeding Behavior; Self-Control

STUDY DESIGN:
Intervention Model Description: Individually randomised, two-arm, parallel-group randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIMISE intervention (Experimental): After a baseline week of self-monitoring their meat consumption, participants will receive health and environmental feedback on their consumption and will be prompted to think about how they could reduce their intake. They will be asked to pre-select strategies from a list of meat consumption reduction actions and set themselves a meat reduction goal.
  During the following four weeks (weeks 2-5), participants will be asked every morning to log their meat consumption of the previous day, plan one of their chosen actions and formulate an if-then plan. Participants will receive weekly feedback on their achieved meat reduction in comparison to week 1.
  After the completion of the fifth week (follow-up 1), participants will be asked to continue performing the actions they found useful for the next four weeks (weeks 6-9). During the ninth week (follow-up 2) participants will be invited back to log their meat intake.
  Interventions: Behavioral: OPTIMISE
- Control (No Intervention): After a baseline week of self-monitoring their meat consumption participants will be asked to try and reduce their meat consumption over the next eight weeks, with no further guidance. They will be invited back to complete log their meat consumption of the previous day during weeks five and nine (follow-up 1 and 2).

INTERVENTIONS:
Behavioral: OPTIMISE — Self-regulation intervention
  Arms: OPTIMISE intervention

SUMMARY:
This randomised controlled trial will test the effectiveness of a self-regulation intervention for reducing meat consumption in people who are motivated to change their meat-eating habits.

DETAILED DESCRIPTION:
An individually randomised, two-arm, parallel-group design will be employed, assessing superiority of the self-regulation intervention over a control. The intervention aims to support individuals in self-monitoring their meat consumption, learning about the impact of their food choices on their health and the environment and setting personal meat reduction goals as well as implementing those goals to reduce meat consumption in manageable steps.

After a baseline week of self-monitoring meat consumption, the intervention will be delivered over four weeks, followed by a four-week long maintenance phase.The study will be delivered remotely through our bespoke website developed specifically for the intervention.

All participants will complete a baseline questionnaire that asks about their demographic characteristics, assesses their self-efficacy regarding consumption of meat-free dishes and asks about their meat-eating identity. Participants will be then randomised 1:1 to the control or intervention group. During the baseline week (week 1, days 2-5), participants will be invited to complete a meat frequency questionnaire, daily, each time looking back at the previous day. After the baseline week, participants will follow their assigned condition for eight weeks. In the control condition, participants will be asked to try and reduce their meat intake, without further guidance. In the intervention condition, participants will be guided through an experimentation process for the first four weeks. This includes setting a meat reduction goal, tracking meat intake daily, planning and implementing an action to reduce meat intake daily and evaluating those actions weekly. After these four weeks (weeks 2-5), intervention group participants will enter a four-week long maintenance phase during which they will be asked to continue with the actions they found useful in the previous weeks. During the fifth and ninth weeks, all participants will be invited to complete the meat frequency questionnaire daily. On the last day of both the fifth and ninth weeks, participants will be asked to complete the self-efficacy and meat-identity questionnaires used in the baseline session again. On the last day of the fifth-week participants of the intervention condition will be further asked to complete a questionnaire to evaluate the intervention. On the last day of the ninth-week participants of the control condition will be asked what kinds of strategies they used to actively reduce their meat intake in the last eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to give informed consent
* Be resident in the UK
* Self report to speak English fluently
* Self-report to eat meat at least five times per week
* Be willing to reduce their meat intake
* Have access to devices compatible with the delivery format of the intervention

Exclusion Criteria:

* Enrolled in another dietary intervention study
* Trying to lose weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Change in mean daily meat consumption from baseline to follow-up 1, comparing intervention and control groups. | five weeks
  Meat consumption was measured with meat-frequency questionnaires administered daily during the baseline week and follow-up 1.

SECONDARY OUTCOMES:
Change in mean daily meat consumption from baseline to follow-up 2, comparing intervention and control groups. | nine weeks
  Meat consumption was measured with meat-frequency questionnaires administered daily during the baseline week and follow-up 2.
Change in mean daily meat consumption from follow-up 1 to follow-up 2, comparing intervention and control groups. | nine weeks
  Meat consumption was measured with meat-frequency questionnaires administered daily during follow-up 1 and follow-up 2.
Change in mean daily consumption of meat subgroups from baseline to both follow-ups, comparing intervention and control groups. | five and nine weeks
  Meat subgroups assessed: red meat, processed meat, and red & processed meat.
Change in meat-free self-efficacy from baseline to both follow-ups, comparing intervention and control groups. | five and nine weeks
  Self-efficacy was measured using three items from the self-efficacy scale Lacroix & Gifford (2019):
  "I lack the cooking skills to prepare meat-free meals" "I don't know what to eat instead of meat" "I don't have enough willpower to not eat meat"
  Answers were given on a 7-point Likert scale ranging from (1) "strongly disagree" to 7 "strongly agree".
Change in participants meat-eating identity from baseline to both follow-ups, comparing intervention and control groups. | five and nine weeks
  Meat identity questionnaire was used to categorise people as follows: 1) meat-eating identity, 2) reduced meat-eating identity, and 3) non-meat eating identity.
  Participants who moved from 1 to 2, 1 to 3, or 2 to 3 were coded as positive meat-identity change=1 and other changes/no change were coded as positive meat-identity change=0
Comparison of actions taken by the control group participants and those taken by the intervention group. | nine weeks
  Control group participants completed a questionnaire at follow-up 2 which asked what strategies they had tried to reduce their meat consumption. Reponses were free-text and explored qualitatively. We assessed which meat reduction actions were chosen by our intervention group participants and compared these to those reported by the control group.
Acceptability of the self-regulation intervention for reducing meat consumption | five weeks
  Acceptability was assessed with an intervention evaluation questionnaire administered at follow-up 1 to intervention group participants.
  The questionnaire asked participants to rate the usefulness of individual intervention components (tracking meat consumption daily, health/environmental feedback, action planning) and additional resources (weekly action evaluation, downloadable action diary, downloadable action overview, links to other resources, ability to review your journey) on a scale of 1 (not useful) to 10 (very useful). We also asked if participants had any additional feedback - this was a free-text question and responses were coded and analysed qualitatively.
Percentage of meat frequency questionnaires completed by participants | nine weeks
  Intervention group participants could complete a maximum of 42 meat frequency questionnaires (daily weeks 1-5 and 9) over the study period, while control group participants could complete a maximum of 21 meat frequency questionnaires (daily weeks 1, 5 and 9). For each participant we calculated their percentage of meat frequency questionnaires submitted (i.e. X/42* 100 or X/21* 100).
  We then looked at the percentage of participants who completed all sessions, and at least 80% of sessions, in both groups.

OTHER OUTCOMES:
Outlier sensitivity analysis of primary outcome | five weeks
  We ran a sensitivity analysis repeating the primary analysis (change in mean daily meat consumption from baseline to follow-up 1) excluding days in which participant total meat intake exceeded 1.5 kg (measured by the meat frequency questionnaires) to assess the effect of outliers.
Barriers to adherence to meat reduction actions | five weeks
  Barriers were identified by open-text responses to daily (Weeks 2-5) action completion question when participants indicated they didn't stick to their action: "Please tell us a little bit more about why you were unable to stick to the action you had planned."

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Jebb, PhD, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Department of Primary Care Health Sciences, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. All data is anonymous at the time of collection.

REFERENCES:
- [Derived] Frie K, Stewart C, Piernas C, Cook B, Jebb SA. Effectiveness of an Online Programme to Tackle Individual's Meat Intake through SElf-regulation (OPTIMISE): A randomised controlled trial. Eur J Nutr. 2022 Aug;61(5):2615-2626. doi: 10.1007/s00394-022-02828-9. Epub 2022 Mar 4. PMID 35244757
- See also: Pre-published statistical analysis plan — https://osf.io/4m2p5/